CLINICAL TRIAL: NCT05398120
Title: Testing the Feasibility of a Skills Group for Adolescents and Young Adults at Clinical High-risk for Psychosis
Brief Title: Skills Group for Youth at Clinical High-Risk for Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Horton, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21120012; 1 H79 SM081196-01 (Other Grant/Funding Number: Substance Abuse and Mental Health Services Administration (SAMHSA),PA State Dept/Public Welfare)
Record Dates: First submitted 2022-05-15; First posted 2022-05-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Clinical High-Risk; Psychological
Keywords: Group intervention; Dialectical behavioral therapy skills; Cognitive behavioral therapy skills; Psychosis-risk

STUDY DESIGN:
Intervention Model Description: Participants already receiving services in the psychosis-risk clinic at the University of Pittsburgh will be asked to participate in the psychosis-risk skills group. Data collected on feasibility and outcome measures will occur pre (within 1 month) -post (up to 4-5 months) and half-way (up to 2-3 months) through the intervention.
Masking Description: There is one condition so masking is not relevant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skills Group (Experimental): There will be one condition which is the group and participants will complete feasibility and outcome measures at baseline, at midpoint, and at the end of the group.
  Interventions: Behavioral: Skills Group

INTERVENTIONS:
Behavioral: Skills Group — Adolescents and young adults with a CHR syndrome ages 13-18 will complete feasibility and outcome measures while participating in a weekly skills group for 6 months.
  Other Names: Psychosis-risk skills group

SUMMARY:
This study is intended to test the feasibility of an integrated cognitive behavioral therapy (CBT) and dialectical behavioral therapy (DBT) skills group for adolescents and young adults at clinical high-risk (CHR) for psychosis. The current study applies a skills group drawing from evidence-based practices (e.g., cognitive behavioral therapy (CBT), dialectical behavioral therapy (DBT)) to those at CHR for psychosis. Up to 30 CHR individuals (starting with a minimum of 3 participants, N accounts for attrition as well), aged 13-18, already receiving clinical services within the HOPE team at University of Pittsburgh will be offered a weekly skills group. Data collected on feasibility and outcome measures will occur pre (within 1 month) -post (up to 4-5 months) and half-way (up to 2-3 months) through the intervention. Taken together, the aim of the proposed intervention is to provide novel insights regarding the utility of a newly developed intervention that integrates both CBT and DBT skills for those at CHR for psychosis.

DETAILED DESCRIPTION:
The goal of the current study is to integrate cognitive behavioral therapy and dialectical behavioral therapy skills and implement in a group format to a sample of individuals at risk for developing a psychotic disorder. These data have the potential to provide a foundation for intervention development in this area. The group will include weekly sessions for 90 minutes with up to 8 members in the group at a time. Each session will include mindfulness, homework review, and skill development. Each individual in the group will be asked to complete the group for 15-weeks. In the first section of the group, skills will be taught to manage and reduce stress. The second set of skills will include teaching individuals how to improve self-disturbances. The final section of the group will include helping participants improve social skills. Furthermore, parents will be asked to participate in a parent/guardian session 1x a month and will also be asked to also fill out a post-group surveys although this is not mandatory.

It is important to note that all hypotheses are exploratory given the feasibility nature of this study and the sample size. Even so, it is predicted, in an exploratory fashion, that this group will be feasible to implement and there will be improvements in symptoms and functioning.

Changes have been made starting Nov 2024 to the group given the feedback received: (1) Instead of 21-weeks, the group has been modified to to 15-weeks, (2) skills are consistent across stages, implementing only standard DBT skills (instead of radically-open DBT: this applies to stage 3 of the group where the goal is intended to improve social impairments), and (3) the number of outcome measures have been reduced and streamlined to follow the general clinic assessment battery to reduce participant burden.

ELIGIBILITY:
Participant Inclusion Criteria:

* 13-18 years of age
* Meet criteria for clinical high-risk syndrome (i.e., at clinical high risk for developing a psychotic disorder). CHR status is determined based off of scoring a 3 (moderate) - 5 (severe) on the Structured Interview for Psychosis-Risk Syndromes and/or having a first degree relative with psychotic disorder and/or the individual meets criteria for schizotypal personality disorder. Additionally individuals with a brief intermittent psychotic symptoms can be included as well (e.g., frankly psychotic symptoms that are very brief)
* Individuals must be enrolled in the HOPE team at the University of Pittsburgh since this group is embedded within that service

Participation Exclusion Criteria:

* Group member meeting criteria for a current/past psychotic disorder

Inclusion Criteria for Parents or Legal Guardians:

* Must be the parent, legal guardian of a 13-18 year-old
* For parents of CHR adolescents, their adolescent must meet criteria for a psychosis-risk syndrome

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Attrition | Up to 5 months
  Feasibility measure; this will be assessed by recording the number of individuals that discontinued group participation.
Attendance | Up to 5 months
  Feasibility measure; daily attendance will be recorded.
Modified Quick Lecomte and Leclerc Scale | Up to 5 months
  Feasibility measure; this modified measure is a a 15-item feasibility measure that assesses feelings about the relevance and importance of group, alliance with the therapists, the group cohesion, appreciation of the group therapy, optimism for the future (five items), feelings about self and others (two items), current mood/anxiety (seven items), distressing thoughts (one item), and feelings about meeting goals (one item). The measure collects data on a 3-point likert scale (0-2), with higher score indicating more group satisfaction/improvement. A mean total score will be collected for each dimension and can range from 0-2. An improvement score taking the proportion of better than usual compared to worse than usual can be calculated for each month of therapy as well.
Participation Scale | Up to 5 months
  Feasibility measure; this is a 9-item checklist assessing the participation and behavior of each group member, with each item rated on a 0 (absence of behavior) to 4 (strong presence of behavior) scale. A total score is computed for each person (range 0-36 scale), as well as an average for all group members, with higher scores indicating more group engagement and prosocial behaviors.
Change from baseline in the participant group survey at up to 3 months | Baseline vs. up to 3 months
  Feasibility measure; this includes 3 questions about the goals for group and asks general questions about how different areas of the individual's life is going (e.g., feeling present, coping with stress, feeling towards self, 10 questions ranging from 0-40) - individuals are to answer on a 0 (much worse) to 4 (greatly improved) scale with higher scores signaling more improvement. Furthermore, this questionnaire also includes questions about the quality of the group from the participants perspective which will provide qualitative data.
Change from up to 3 months in the participant group survey at up to 5 months | Up to 3 months vs up to 5 months
  Feasibility measure; this includes 3 questions about the goals for group and asks general questions about how different areas of the individual's life is going (e.g., feeling present, coping with stress, feeling towards self, 10 questions ranging from 0-40) - individuals are to answer on a 0 (much worse) to 4 (greatly improved) scale with higher scores signaling more improvement. Furthermore, this questionnaire also includes questions about the quality of the group from the participants perspective which will provide qualitative data.
Change from baseline in the participant group survey at up to 5 months | Baseline vs. up to 5 months
  Feasibility measure; this includes 3 questions about the goals for group and asks general questions about how different areas of the individual's life is going (e.g., feeling present, coping with stress, feeling towards self, 10 questions ranging from 0-40) - individuals are to answer on a 0 (much worse) to 4 (greatly improved) scale with higher scores signaling more improvement. Furthermore, this questionnaire also includes questions about the quality of the group from the participants perspective which will provide qualitative data.
Change from baseline in Satisfaction with Therapy and Therapist Scale at up to 3 months | Baseline vs. up to 3 months
  A satisfaction 13-item scale that asks the individual to indicate their level of satisfaction of the therapy and therapists in the group treatment. Scores fall on a 1 (strong disagree) to 5 (strongly agree) scale with higher numbers indicating higher satisfaction. Scores range from 12-60. There is an additional item that falls on a 1-5 scale that asks about how the tre (atment helped with the specific problem that led to therapy, with higher scores indicating that therapy made things worse (range is 1-5).
Change from 3 months in Satisfaction with Therapy and Therapist Scale at up to 5 months | Up to 3 months vs. up to 5 months.
  A satisfaction 13-item scale that asks the individual to indicate their level of satisfaction of the therapy and therapists in the group treatment. Scores fall on a 1 (strong disagree) to 5 (strongly agree) scale with higher numbers indicating higher satisfaction. Scores range from 12-60. There is an additional item that falls on a 1-5 scale that asks about how the tre (atment helped with the specific problem that led to therapy, with higher scores indicating that therapy made things worse (range is 1-5).
Fidelity scores | Up to 5 months
  Fidelity scores developed specifically for this group asking questions about the structure of the group meant to be filled out by co-leaders (e.g., was there a mindfulness practice in the session?). Each item can have a Yes or No response. More Yes responses indicate more fidelity. There are a total of 9 items.

SECONDARY OUTCOMES:
Change from baseline in Lehman Quality of Life Functional Assessment at up to 3 months. | Baseline vs. up to 3 months
  A brief 4- item questionnaire that asks about general feelings about one's life, the amount of fun in life, feeling towards others, and amount of time spent with others on a scale of 0 (terrible) to 6 (delightful) scale. Scores range from 0-24, with lower scores indicating lower quality of life. ~2 minutes
Change from up to 3 months in Lehman Quality of Life Functional Assessment at up to 5 months. | Up to 3 months vs. up to 5 months
  A brief 4- item questionnaire that asks about general feelings about one's life, the amount of fun in life, feeling towards others, and amount of time spent with others on a scale of 0 (terrible) to 6 (delightful) scale. Scores range from 0-24, with lower scores indicating lower quality of life. ~2 minutes
Change from baseline in Lehman Quality of Life Functional Assessment at up to 5 months. | Baseline vs. up to 5 months
  A brief 4- item questionnaire that asks about general feelings about one's life, the amount of fun in life, feeling towards others, and amount of time spent with others on a scale of 0 (terrible) to 6 (delightful) scale. Scores range from 0-24, with lower scores indicating lower quality of life. ~2 minutes
Change from baseline in Perceived Stress Scale at up to 3 months | Baseline to up to 3 months
  A 10-item questionnaire that measures the degree to which situations in one's life are appraised as stressful. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives. Some items are reversed scored. Ratings are collected on a 0 ("never") to 4 ("very often") scale with higher scores indicating more perceived stress, range is 0-40.
Change from up to 3 months in Perceived Stress Scale at up to 5 months. | Up to 3 months vs. up to 5 months
  A 10-item questionnaire that measures the degree to which situations in one's life are appraised as stressful. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives. Ratings are collected on a 0 ("never") to 4 ("very often") scale with higher scores indicating more perceived stress, range is 0-40.
Change from baseline in Perceived Stress Scale at up to 5 months. | Baseline to up to 5 months
  A 10-item questionnaire that measures the degree to which situations in one's life are appraised as stressful. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives. Ratings are collected on a 0 ("never") to 4 ("very often") scale with higher scores indicating more perceived stress, range is 0-40.
Change from baseline in Cognitive Insight Scale at up to 3 months | Baseline vs. up to 3 months
  A 15-item measure evaluating patient's self-reflectiveness and their overconfidence in their interpretations of their experiences. Ratings are collected on a 0 "do not agree at all" to 3 "agree completely" scale ranging from 0-45. A 9-item self-reflectiveness subscale (range 0-27) and a 6-item self-certainty subscale (range 0-18) are also made. Higher scores indicate more insight, self-reflectiveness, and more self-certainty. A composite index of the insight reflecting cognitive insight is calculated by subtracting the score for the self-certainty scale from that of the self-reflectiveness scale where lower numbers indicate less insight.
Change from up to 3 months in Cognitive Insight Scale at up to 5 months. | Up to 3 months vs. up to 5 months
  A 15-item measure evaluating patient's self-reflectiveness and their overconfidence in their interpretations of their experiences. Ratings are collected on a 0 "do not agree at all" to 3 "agree completely" scale ranging from 0-45. A 9-item self-reflectiveness subscale (range 0-27) and a 6-item self-certainty subscale (range 0-18) are also made. Higher scores indicate more insight, self-reflectiveness, and more self-certainty. A composite index of the insight reflecting cognitive insight is calculated by subtracting the score for the self-certainty scale from that of the self-reflectiveness scale where lower numbers indicate less insight.
Change from baseline in Cognitive Insight Scale at up to 5 months. | Baseline vs. up to 5 months
  A 15-item measure evaluating patient's self-reflectiveness and their overconfidence in their interpretations of their experiences. Ratings are collected on a 0 "do not agree at all" to 3 "agree completely" scale ranging from 0-45. A 9-item self-reflectiveness subscale (range 0-27) and a 6-item self-certainty subscale (range 0-18) are also made. Higher scores indicate more insight, self-reflectiveness, and more self-certainty. A composite index of the insight reflecting cognitive insight is calculated by subtracting the score for the self-certainty scale from that of the self-reflectiveness scale where lower numbers indicate less insight.
Change from baseline in Defeatist Performance Attitudes at up to 3 months | Baseline vs. Up to 3 months
  A 15-item questionnaire assessing dysfunctional attitudes commonly targeted by CBT therapy. Items are rated on a 1-7 Likert scale and higher total scores (range = 15-105) indicate more severe defeatist performance attitudes.
Change from up to 3 months in Defeatist Performance Attitudes at up to 5 months. | Up to 3 months vs up to 5 months
  A 15-item questionnaire assessing dysfunctional attitudes commonly targeted by CBT therapy. Items are rated on a 1-7 Likert scale and higher total scores (range = 15-105) indicate more severe defeatist performance attitudes.
Change from baseline in Defeatist Performance Attitudes at up to 5 months. | Baseline vs. up to 5 months
  A 15-item questionnaire assessing dysfunctional attitudes commonly targeted by CBT therapy. Items are rated on a 1-7 Likert scale and higher total scores (range = 15-105) indicate more severe defeatist performance attitudes.
Change from baseline in Avoidance Fusion Questionnaire for Youth at up to 3 months | Baseline vs. up to 3 months
  17 items assessing psychological acceptance on a 1 (not at all true) to 5 (very true) scale. Sum scores can range from 17-85 with higher scores representing more psychological inflexibility.
Change from up to 3 months in Avoidance Fusion Questionnaire for Youth at up to 5 months | Up to 3 months vs. up to 5 months
  17 items assessing psychological acceptance on a 1 (not at all true) to 5 (very true) scale. Sum scores can range from 17-85 with higher scores representing more psychological inflexibility.
Change from baseline in Avoidance Fusion Questionnaire for Youth at up to 5 months | Baseline vs. up to 5 months
  17 items assessing psychological acceptance on a 1 (not at all true) to 5 (very true) scale. Sum scores can range from 17-85 with higher scores representing more psychological inflexibility.
Change from baseline in Social and Role Functioning Scale at up to 3 months | Baseline vs. up to 3 months
  A brief interview assessing social and role areas of functioning not confounded by symptom ratings and appropriate across life spans; high scores indicate better social functioning. Scores fall on a 1-10 scale.
Change from up to 3 months in Social and Role Functioning Scale at up to 5 months | Up to 3 months vs. up to 5 months
  A brief interview assessing social and role areas of functioning not confounded by symptom ratings and appropriate across life spans; high scores indicate better social functioning. Scores fall on a 1-10 scale.
Change from baseline in Social and Role Functioning Scale at up to 5 months | Baseline vs. up to 5 months
  A brief interview assessing social and role areas of functioning not confounded by symptom ratings and appropriate across life spans; high scores indicate better social functioning. Scores fall on a 1-10 scale.
Change in symptoms from baseline Structured Interview for Psychosis-Risk Syndromes and/or Mini interview (abbreviated version) to up to 3 months | Baseline vs. up to 3 months
  An interview designed to assess five domains of positive symptoms (e.g., seeing shadows). Ratings are given by assessors on a 0 (absent) to 6 (severe) scale. Higher ratings indicate more symptom severity. Scores range from 0-30.
Change from up to 3 months on the Structured Interview for Psychosis-Risk Syndromes interview and/or Mini interview (abbreviated version) at up to 5 months | Up to 3 months vs. up to 5 months
  An interview designed to assess five domains of positive symptoms (e.g., seeing shadows). Ratings are given by assessors on a 0 (absent) to 6 (severe) scale. Higher ratings indicate more symptom severity. Scores range from 0-30.
Change from baseline in the Structured Interview for Psychosis-Risk Syndromes interview and/or Mini interview (abbreviated version) at up to 5 months | Baseline vs. up to 5 months
  An interview designed to assess five domains of positive symptoms (e.g., seeing shadows). Ratings are given by assessors on a 0 (absent) to 6 (severe) scale. Higher ratings indicate more symptom severity. Scores range from 0-30.
Change from baseline in Negative Symptom Inventory Psychosis-Risk at up to 3 months | Baseline vs. up to 3 months
  A brief, 11-item assessment of negative symptoms, with higher scores indicating more negative symptoms. Two items assess avolition (i.e., reduced motivational behavior and experience), three items assess asociality (i.e., reduction in the desire for and engagement in social activities), two items assess anhedonia (i.e., reduction in pleasure in activities), three items related to affect, and 1 related to quantity of speech. Each of these subscales are summed and/or averaged and there is a total score (range is 0-55) with higher scores indicating more negative symptom severity.
Change from up to 3 months in Negative Symptom Inventory Psychosis-Risk at up to 5 months | Up to 3 months vs. up to 5 months
  A brief, 11-item assessment of negative symptoms, with higher scores indicating more negative symptoms. Two items assess avolition (i.e., reduced motivational behavior and experience), three items assess asociality (i.e., reduction in the desire for and engagement in social activities), two items assess anhedonia (i.e., reduction in pleasure in activities), three items related to affect, and 1 related to quantity of speech. Each of these subscales are summed and/or averaged and there is a total score (range is 0-55) with higher scores indicating more negative symptom severity.
Change from baseline in Negative Symptom Inventory Psychosis-Risk at up to 5 months | Baseline vs. up to 5 months
  A brief, 11-item assessment of negative symptoms, with higher scores indicating more negative symptoms. Two items assess avolition (i.e., reduced motivational behavior and experience), three items assess asociality (i.e., reduction in the desire for and engagement in social activities), two items assess anhedonia (i.e., reduction in pleasure in activities), three items related to affect, and 1 related to quantity of speech. Each of these subscales are summed and/or averaged and there is a total score (range is 0-55) with higher scores indicating more negative symptom severity.
Change from baseline in Beck Depression Inventory to up to 3 months | Baseline vs. up to 3 months
  A 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression on a 4 point likert scale with higher scores indicating more depressive symptoms, range 0-63.
Change from up to 3 months in Beck Depression Inventory to up to 5 months | Up to 3 months vs. up to 5 months
  A 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression on a 4 point likert scale with higher scores indicating more depressive symptoms, range 0-63.
Change from baseline in Beck Depression Inventory to up to 5 months | Baseline vs. up to 5 months
  A 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression on a 4 point likert scale with higher scores indicating more depressive symptoms, range 0-63.
Change from baseline in Beck Anxiety Inventory at up to 3 months | Baseline vs. up to 3 months
  A 21-item scale measuring common symptoms of anxiety on a 4 point likert scale with higher scores indicating more anxiety, range 0-63.
Change from up to 3 months in Beck Anxiety Inventory at up to 5 months | Up to 3 months vs. up to 5 months
  A 21-item scale measuring common symptoms of anxiety on a 4 point likert scale with higher scores indicating more anxiety, range 0-63.
Change from baseline in Beck Anxiety Inventory at up to 5 months | Baseline vs. up to 5 months
  A 21-item scale measuring common symptoms of anxiety on a 4 point likert scale with higher scores indicating more anxiety, range 0-63.
Child Trauma Questionnaire | Baseline
  A 28-item screen designed to assess the degree to which different traumatic experiences apply to the individual (e.g., never true (1), rarely (2), sometimes true (3), often true (4), very often true (5)). Higher total scores indicate more traumatic events and scores can range from 28-140. Some items are reverse scored. This questionnaire also measures subscales that have five items each: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Each subscale ranges from 5-25 with higher scores indicating more trauma exposure.
Change from baseline Child and Adolescent Mindfulness Measure at up to 3 months | Baseline vs. up to 3 months
  A 10 item measure that assesses present-moment awareness and nonjudgmental, nonavoidant responses to thoughts and feelings. Ratings are collected on a 0 (never true) to 4 (always true) and are reverse scored. Scores range from 0-40. Higher scores indicate higher levels of mindfulness.
Change from up to 3 months Child and Adolescent Mindfulness Measure at up to 5 months | up to 3 months vs. up to 5 months
  A 10 item measure that assesses present-moment awareness and nonjudgmental, nonavoidant responses to thoughts and feelings. Ratings are collected on a 0 (never true) to 4 (always true) and are reverse scored. Scores range from 0-40. Higher scores indicate higher levels of mindfulness.
Change from baseline Child and Adolescent Mindfulness Measure at up to 5 months | Baseline vs. up to 5 months
  A 10 item measure that assesses present-moment awareness and nonjudgmental, nonavoidant responses to thoughts and feelings. Ratings are collected on a 0 (never true) to 4 (always true) and are reverse scored. Scores range from 0-40. Higher scores indicate higher levels of mindfulness.
Change from baseline in Emotion Regulation Questionnaire at up to 3 months | Baseline vs. up to 3 months
  A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree), and higher scores indicate more use of the noted strategies. Cognitive reappraisal (six items, range 6-42) and expressive suppression items (four items, range 4-28).
Change from up to 3 months in Emotion Regulation Questionnaire at up to 5 months | Up to 3 months vs. up to 5 months
  A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree), and higher scores indicate more use of the noted strategies. Cognitive reappraisal (six items, range 6-42) and expressive suppression items (four items, range 4-28).
Change from baseline in Emotion Regulation Questionnaire at up to 5 months | Baseline vs. up to 5 months
  A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree), and higher scores indicate more use of the noted strategies. Cognitive reappraisal (six items, range 6-42) and expressive suppression items (four items, range 4-28).
Change from baseline in Social Connectedness Scale at up to 3 months | Baseline vs. up to 3 months
  A 20-item measure to assess how connected one feels to others in their social environment on a 1 (strongly disagree to 6 (strongly agree) scale. All of the items are reversed and are then summed for a total score. A high score reflects more connectedness, range is 20-120.
Change from up to 3 months in Social Connectedness Scale at up to 5 months | Up to 3 months vs. up to 5 months
  A 20-item measure to assess how connected one feels to others in their social environment on a 1 (strongly disagree to 6 (strongly agree) scale. All of the items are reversed and are then summed for a total score. A high score reflects more connectedness, range is 20-120.
Change from baseline in Social Connectedness Scale at up to 5 months | Baseline vs. up to 5 months
  A 20-item measure to assess how connected one feels to others in their social environment on a 1 (strongly disagree to 6 (strongly agree) scale. All of the items are reversed and are then summed for a total score. A high score reflects more connectedness, range is 20-120.
Change in Internalized Stigma Mental Illness Inventory (ISMI) baseline up to 3 months | Baseline vs. up to 3 months
  A 29 item measure that assesses self-stigma on a 1 (strong disagree) - 4 (strongly agree) scale. Scores can range from 29-116 with higher scores indicating more self-stigma. Subscales include alienation, stereotype endorsement, perceived discrimination, social withdrawal, and stigma resistance.
Change in Internalized Stigma Mental Illness Inventory (ISMI) from up to 3 months to up to 5 months | Up to 3 months vs. up to 5 months
  A 29 item measure that assesses self-stigma on a 1 (strong disagree) - 4 (strongly agree) scale. Scores can range from 29-116 with higher scores indicating more self-stigma. Subscales include alienation, stereotype endorsement, perceived discrimination, social withdrawal, and stigma resistance.
Change in Internalized Stigma Mental Illness Inventory (ISMI) baseline up to 5 months | Baseline vs. up to 5 months
  A 29 item measure that assesses self-stigma on a 1 (strong disagree) - 4 (strongly agree) scale. Scores can range from 29-116 with higher scores indicating more self-stigma. Subscales include alienation, stereotype endorsement, perceived discrimination, social withdrawal, and stigma resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Horton, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Bellefield Towers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying publication will be shared including data dictionaries after publication and in line with the grantee policies regarding data sharing. Data will be de-identified before sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Data sharing will be occur when specific requests to analyze data are made by investigators in the field and in line with grant funder data sharing policies

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Cane, D.B. Olinger, L.J,. Gotlib, I.H., Kuiper, N.A. (1986) Factor structure of the Dysfunctional Attitude Scale in a student population. J Clin Psychol. 42, 307 - 309 .
- [Background] Benedict, R. H. B., Schretlen, D., Groninger, L., & Brandt, J. (1998). The Hopkins verbal learning test-revised: Normative data and analysis of interform and test-retest reliability. Clinical Neuropsychologist, 12, 43-55.
- [Background] Keefe RS, Goldberg TE, Harvey PD, Gold JM, Poe MP, Coughenour L. The Brief Assessment of Cognition in Schizophrenia: reliability, sensitivity, and comparison with a standard neurocognitive battery. Schizophr Res. 2004 Jun 1;68(2-3):283-97. doi: 10.1016/j.schres.2003.09.011. PMID 15099610
- [Background] Greco LA, Lambert W, Baer RA. Psychological inflexibility in childhood and adolescence: development and evaluation of the Avoidance and Fusion Questionnaire for Youth. Psychol Assess. 2008 Jun;20(2):93-102. doi: 10.1037/1040-3590.20.2.93. PMID 18557686
- [Background] Cornblatt BA, Auther AM, Niendam T, Smith CW, Zinberg J, Bearden CE, Cannon TD. Preliminary findings for two new measures of social and role functioning in the prodromal phase of schizophrenia. Schizophr Bull. 2007 May;33(3):688-702. doi: 10.1093/schbul/sbm029. Epub 2007 Apr 17. PMID 17440198
- [Background] Lee, R. M., & Robbins, S. B. (1995). Measuring belongingness: The Social Connectedness and the Social Assurance Scales. Journal of Counseling Psychology, 42, 232-241.
- [Background] Miller TJ, McGlashan TH, Woods SW, Stein K, Driesen N, Corcoran CM, Hoffman R, Davidson L. Symptom assessment in schizophrenic prodromal states. Psychiatr Q. 1999 Winter;70(4):273-87. doi: 10.1023/a:1022034115078. PMID 10587984
- [Background] Loewy RL, Pearson R, Vinogradov S, Bearden CE, Cannon TD. Psychosis risk screening with the Prodromal Questionnaire--brief version (PQ-B). Schizophr Res. 2011 Jun;129(1):42-6. doi: 10.1016/j.schres.2011.03.029. Epub 2011 Apr 20. PMID 21511440
- [Background] McGlashan, T. H., Walsh, B. C., Woods, S. W., Addington, J., Cadenhead, K., Cannon, T., & Walker, E. (2001). Structured interview for psychosis-risk syndromes. New Haven, CT: Yale School of Medicine.
- [Background] Pelletier-Baldelli A, Strauss GP, Visser KH, Mittal VA. Initial development and preliminary psychometric properties of the Prodromal Inventory of Negative Symptoms (PINS). Schizophr Res. 2017 Nov;189:43-49. doi: 10.1016/j.schres.2017.01.055. Epub 2017 Feb 8. PMID 28189529
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Kenardy JA, Spence SH, Macleod AC. Screening for posttraumatic stress disorder in children after accidental injury. Pediatrics. 2006 Sep;118(3):1002-9. doi: 10.1542/peds.2006-0406. PMID 16950991
- [Background] Bernstein, D., & Fink, L. (1998). Childhood Trauma Questionnaire: A retrospective self-report. San Antonio, TX: The Psychological Corporation.
- [Background] Lynch, T. R. (2018b). Radically Open Dialectical Behavior Therapy: Theory and practice for treating disorders of overcontrol. Reno, NV: Context Press, an imprint of New Harbinger Publications, Inc.
- [Background] Greco LA, Baer RA, Smith GT. Assessing mindfulness in children and adolescents: development and validation of the Child and Adolescent Mindfulness Measure (CAMM). Psychol Assess. 2011 Sep;23(3):606-14. doi: 10.1037/a0022819. PMID 21480722
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Lecomte, T., Leclerc, C. & Wykes, T. 2003. Quick LL. Group CBT for Psychosis: A Guidebook for Clinicians.
- [Background] Fusar-Poli P, Borgwardt S, Bechdolf A, Addington J, Riecher-Rossler A, Schultze-Lutter F, Keshavan M, Wood S, Ruhrmann S, Seidman LJ, Valmaggia L, Cannon T, Velthorst E, De Haan L, Cornblatt B, Bonoldi I, Birchwood M, McGlashan T, Carpenter W, McGorry P, Klosterkotter J, McGuire P, Yung A. The psychosis high-risk state: a comprehensive state-of-the-art review. JAMA Psychiatry. 2013 Jan;70(1):107-20. doi: 10.1001/jamapsychiatry.2013.269. PMID 23165428
- [Background] Lynch TR, Hempel RJ, Dunkley C. Radically Open-Dialectical Behavior Therapy for Disorders of Over-Control: Signaling Matters. Am J Psychother. 2015;69(2):141-62. doi: 10.1176/appi.psychotherapy.2015.69.2.141. PMID 26160620
- [Background] McCauley E, Berk MS, Asarnow JR, Adrian M, Cohen J, Korslund K, Avina C, Hughes J, Harned M, Gallop R, Linehan MM. Efficacy of Dialectical Behavior Therapy for Adolescents at High Risk for Suicide: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Aug 1;75(8):777-785. doi: 10.1001/jamapsychiatry.2018.1109. PMID 29926087
- [Background] Linehan MM, Korslund KE, Harned MS, Gallop RJ, Lungu A, Neacsiu AD, McDavid J, Comtois KA, Murray-Gregory AM. Dialectical behavior therapy for high suicide risk in individuals with borderline personality disorder: a randomized clinical trial and component analysis. JAMA Psychiatry. 2015 May;72(5):475-82. doi: 10.1001/jamapsychiatry.2014.3039. PMID 25806661
- [Background] Strauss GP, Pelletier-Baldelli A, Visser KF, Walker EF, Mittal VA. A review of negative symptom assessment strategies in youth at clinical high-risk for psychosis. Schizophr Res. 2020 Aug;222:104-112. doi: 10.1016/j.schres.2020.04.019. Epub 2020 Jun 7. PMID 32522469
- [Background] Lenz, A.S., James, P., Stewart, C. et al. A Preliminary Validation of the Youth Over- and Under-Control (YOU-C) Screening Measure with a Community Sample. Int J Adv Counselling 43, 489-503 (2021). https://doi.org/10.1007/s10447-021-09439-9
- [Background] Lehman, A., Kernan, E., & Postrado, L.Toolkit Evaluating Quality of Life for Persons with Severe Mental Illness. https://www.hsri.org/publication/toolkit_evaluating_quality_of_life_for_persons_with_severe_mental_illn
- [Background] Lehman, A.F. (1988). A quality of life interview for the chronically mentally ill. Evaluation and Program Planning, 11, 51-62.
- [Background] Oei, Tian Po & Green, Angela. (2008). The Satisfaction With Therapy and Therapist Scale-Revised (STTS-R) for Group Psychotherapy: Psychometric Properties and Confirmatory Factor Analysis. Professional Psychology Research and Practice. 39. 10.1037/0735-7028.39.4.435.
- [Background] Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: psychometric properties of a new measure. Psychiatry Res. 2003 Nov 1;121(1):31-49. doi: 10.1016/j.psychres.2003.08.008. PMID 14572622
- [Background] Woods SW, Lympus C, McGlashan TH, Walsh BC, Cannon TD. The Mini-SIPS: development of a brief clinical structured interview guide to diagnosing DSM-5 Attenuated Psychosis Syndrome and training outcomes. BMC Psychiatry. 2022 Dec 13;22(1):784. doi: 10.1186/s12888-022-04406-z. PMID 36514073
- [Derived] Gupta T, Antezana L, Porter C, Mayanil T, Bylsma LM, Maslar M, Horton LE. Skills program for awareness, connectedness, and empowerment: A conceptual framework of a skills group for individuals with a psychosis-risk syndrome. Front Psychiatry. 2023 Mar 2;14:1083368. doi: 10.3389/fpsyt.2023.1083368. eCollection 2023. PMID 37025348